CLINICAL TRIAL: NCT05073744
Title: Analgesic Efficacy and Safety of Nalbuphine Versus Morphine for Perioperative Tumor Ablation: a Randomized, Control, Multicentre Trial
Brief Title: Nalbuphine Versus Morphine for Perioperative Tumor Ablation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Chair, Center of IR and vascular surgery, Department of radiology, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NPRCT001
Record Dates: First submitted 2021-09-06; First posted 2021-10-11 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Nalbuphine Allergy; Ablation; Safety
MeSH Terms: interventions — Nalbuphine; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumor ablation using nalbuphine for pain control and anaesthesia (Experimental): Nalbuphine hydrochloride injection (80mg) plus 0.9% saline are combined into 80 ml self-controlled analgesic pump, which will be run 25minutes before ablation under Electrocardiogram monitoring. Single pressure administration if numerical rating scale≥4 points.
  Interventions: Drug: Nalbuphine
- Tumor ablation using morphine for pain control and anaesthesia (Active Comparator): Morphine hydrochloride injection (80mg) plus 0.9% saline are combined into 80 ml self-controlled analgesic pump, which will be run 25minutes before ablation under Electrocardiogram monitoring. Single pressure administration if numerical rating scale≥4 points.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Nalbuphine — Nalbuphine hydrochloride injection or morphine hydrochloride injection is used for perioperative tumor ablation
  Other Names: Tumor ablation using nalbuphine
  Arms: Tumor ablation using nalbuphine for pain control and anaesthesia
Drug: Morphine — Morphine hydrochloride injection is used for perioperative tumor ablation
  Other Names: Tumor ablation using morphine
  Arms: Tumor ablation using morphine for pain control and anaesthesia

SUMMARY:
This randomized, positive control, multicentre trial is designed to compare the analgesic efficacy and safety of nalbuphine hydrochloride injection and morphine hydrochloride injection for perioperative tumor ablation.

DETAILED DESCRIPTION:
Sedation and analgesia use in tumor ablation is a necessary part of the procedure. However, the optimal medicine for sedation and analgesia for tumor ablation remains controversial. Currently, morphine is a traditional opioid used for pain control and anaesthesia. As no publications have compared the anaesthetic and analgesic effects between nalbuphine and morphine during tumor ablation, this trial aims to compare the analgesic efficacy and safety of nalbuphine and morphine for perioperative tumor ablation. In addition, other endpoints in term of perioperative analgesia indexes, such as ablation time, daily dose, analgesia satisfaction, quality of life, and safety, etc. will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring tumor ablation;
* Voluntarily participate and sign the informed consent.

Exclusion Criteria:

* Allergic to contrast agent, test drug or other ingredients;
* With a history of substance abuse, chronic pain and mental illness;
* Use of any monamine oxidase inhibitor within 14 days prior to randomization;
* Pregnant or breastfeeding;
* Cannot tolerate ablation due to other reasons;
* Cannot express their wishes correctly;
* Poor compliance, unable to complete the trial;
* Have participated in other drug trials within 30 days prior to enrollment;
* Judged by the researcher to be unsuitable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2021-09-05 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Analgesic efficiency | From the begin to 48 hours after procedure
  No. effective cases / No.Total cases * 100%. The numerical rating scale score at the evaluation time point (at rest) ≤3 is considered as effective analgesia.

SECONDARY OUTCOMES:
Pain intensity | From the begin to 48 hours after procedure
  Pain assessment using the numerical rating scale (NRS), which is composed of 11 numbers spaced from 0 to 10, with 0 representing "no pain" and 10 representing "most intense pain". Patients chose 1 number to represent their pain intensity.
Analgesia satisfaction | Up to 4 hours
  Scored using visual analogue scale, a 10 cm long scale, marked with 10 markers, both ends of 0 point and 10 points respectively. Participant and medical care personnel mark the corresponding position on a ruler that represents their satisfaction. A score of 0 represents extremely dissatisfied and a score of 10 represents very satisfied.
Duration of ablation | Up to 4 hours
  Duration of the whole procedure
Postoperative hospital stay | Up to 10 days
  Days from the time of ablation to Discharge time
Rate of continuous ablation without complaining of pain | Up to 4 hours
  No. ablation without complaining of pain cases / No.Total cases * 100%
Average daily dosage | From nalbuphine/morphine use to 48 hours after procedure
  Total dose of nalbuphine or morphine / Total days of analgesia
Health-related quality of life | 7 days after procedure
  Assessed by telephone, using the standard of Quality of Life Question-Core by the European O-Rganization for Reasearch and Treatment of Cancer (EORTC QLQ-C30 scale,Version 3.0). The evaluation of quality of life from a multi-dimensional perspective can better reflect the connotation of quality of life, which has been applied to measure QOL of cancer patients in many countries and regions. A total of 30 questions will be replied with different points. Higher score represents lower quality of life.

OTHER OUTCOMES:
Safety end point | From nalbuphine/morphine use to 48 hours after procedure
  Adverse reactions related with nalbuphine or morphine according to "Common Terminology Criteria for Adverse Events" by "National Cancer Institute" (NCI-CTCAE, version5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (20):
- China (20):
  - Anhui Province Cancer Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangxi Medical University Affiliated Tumor Hospita, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jingmen NO.2People's Hospital, Jingmen, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Lishui Municipal Central Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Other researchers can contact the PI for data.

REFERENCES:
- [Background] Laurent G, Bertaux G, Martel A, Fraison M, Fromentin S, Gonzalez S, Pierre FS, Wolf JE. A randomized clinical trial of continuous flow nitrous oxide and nalbuphine infusion for sedation of patients during radiofrequency atrial flutter ablation. Pacing Clin Electrophysiol. 2006 Apr;29(4):351-7. doi: 10.1111/j.1540-8159.2006.00352.x. PMID 16650261
- [Background] Sun S, Guo Y, Wang T, Huang S. Analgesic Effect Comparison Between Nalbuphine and Sufentanil for Patient-Controlled Intravenous Analgesia After Cesarean Section. Front Pharmacol. 2020 Nov 16;11:574493. doi: 10.3389/fphar.2020.574493. eCollection 2020. PMID 33364949
- [Background] Yu P, Zhang J, Wang J. Nalbuphine for spinal anesthesia: A systematic review and meta-analysis. Pain Pract. 2022 Jan;22(1):91-106. doi: 10.1111/papr.13021. Epub 2021 Jun 2. PMID 33887111
- [Derived] Xue Y, Huang Z, Cheng B, Sun J, Zhu H, Tang Y, Wang X. Analgesic efficacy and safety of nalbuphine versus morphine for perioperative tumor ablation: a randomized, controlled, multicenter trial. Trials. 2022 Oct 22;23(1):887. doi: 10.1186/s13063-022-06825-5. PMID 36273202